CLINICAL TRIAL: NCT00400985
Title: Sensitivity of the InSync Sentry OptiVol Feature for the Prediction of Heart Failure
Acronym: SENSE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: SENSE-HF, V.1, Dec.8, 2004
Record Dates: First submitted 2005-09-13; First posted 2006-11-17 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; Diagnostic; Ambulatory Monitoring; Intrathoracic Impedance
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable Device diagnostics (Other): All enrolled subjects were implanted with a device. Audible Device diagnostics turned on or off
  Interventions: Device: Implantable device: monitoring of intrathoracic impedance using the OptiVol diagnostic tool.

INTERVENTIONS:
Device: Implantable device: monitoring of intrathoracic impedance using the OptiVol diagnostic tool. — SENSE-HF is non randomized trial. Study divided in 3 phases among which the first phase is blinded towards device diagnostic data.

SUMMARY:
The SENSE-HF study is a prospective, observational, international multi-center study prospectively evaluating the sensitivity and positive predictive value of the OptiVol Fluid Trends data in predicting Heart Failure related hospitalizations and health care utilizations associated with signs and/or symptoms of pulmonary congestion, and to define OptiVol clinical guidelines for subject therapy management.

DETAILED DESCRIPTION:
The SENSE-HF study prospectively evaluates the OptiVol feature in the prediction of Heart Failure related events associated with signs and symptoms of pulmonary congestion and in the subject HF therapy management.

The OptiVol feature is based on the measurement of daily intrathoracic impedance values, measurements that can be used to track changes in the subject's thoracic fluid status over time. An Alert warns the patient whenever a programmable threshold has been reached.

The study is divided into three phases.

The first phase is double-blinded and designed to determine the sensitivity and positive predictive value of the OptiVol Fluid Trends data for the detection of Heart Failure related hospitalizations with signs and/or symptoms of pulmonary congestion.

In the second phase of the study, the Alert is turned ON and the positive predictive value of the first OptiVol Patient Alert for the development of signs and/or symptoms of pulmonary congestion will be evaluated.

The third phase of the study allows for remote subject therapy management using the OptiVol Patient Alert. The patient management strategy is then based on the experience gained in the second study phase Physician actions taken in the occurrence of a Patient Alert will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Successfully implanted InSync Sentry device (< 34 days post implant or pocket revision)in the pectoral region;
* At least one HF-related hospitalization that required administration of IV medication (inotropes, nitrates, diuretics) within the last 12 months
* The Subject has a market released, transvenous, high voltage Right Ventricular lead
* The Subject is able to detect a Patient Alert signal

Exclusion Criteria:

* <18 years of age (or under a minimum age required by local law)
* Moderate to severe Chronic Obstructive Pulmonary Disease (COPD)
* Post heart transplant or awaiting heart transplantation
* Primary pulmonary hypertension
* Renal insufficiency requiring dialysis

Amendment to the inclusion criteria (Jul 06):

* Inclusion of patients with Concerto/Virtuoso devices.
* At least one HF-related hospitalization that required administration of IV (or uptitration of the oral medication)(inotropes, nitrates, diuretics)within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2005-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Conraads, Professor, Principal Investigator — UZA, Antwerpen, Belgium; Martin Cowie, Professor, Principal Investigator — Royal Brompton Hospital, London, UK
Locations (2):
- UZA, Antwerp, Belgium
- Royal Brompton, London, United Kingdom

REFERENCES:
- [Background] Yu CM, Wang L, Chau E, Chan RH, Kong SL, Tang MO, Christensen J, Stadler RW, Lau CP. Intrathoracic impedance monitoring in patients with heart failure: correlation with fluid status and feasibility of early warning preceding hospitalization. Circulation. 2005 Aug 9;112(6):841-8. doi: 10.1161/CIRCULATIONAHA.104.492207. Epub 2005 Aug 1. PMID 16061743
- [Result] Conraads VM, Tavazzi L, Santini M, Oliva F, Gerritse B, Yu CM, Cowie MR. Sensitivity and positive predictive value of implantable intrathoracic impedance monitoring as a predictor of heart failure hospitalizations: the SENSE-HF trial. Eur Heart J. 2011 Sep;32(18):2266-73. doi: 10.1093/eurheartj/ehr050. Epub 2011 Feb 28. PMID 21362703
- [Derived] Conraads VM, Spruit MA, Braunschweig F, Cowie MR, Tavazzi L, Borggrefe M, Hill MR, Jacobs S, Gerritse B, van Veldhuisen DJ. Physical activity measured with implanted devices predicts patient outcome in chronic heart failure. Circ Heart Fail. 2014 Mar 1;7(2):279-87. doi: 10.1161/CIRCHEARTFAILURE.113.000883. Epub 2014 Feb 11. PMID 24519908
- See also: Public website — http://www.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 501 patients from 41 medical clinics in 13 countries were enrolled between March 4, 2005 and September 9, 2008.
Groups:
- All Patients: All study participants received the same treatment
Period: Overall Study
Arm/Group | All Patients
Started | 501
Completed | 449
Not Completed | 52
Not completed — Withdrawal by Subject | 5
Not completed — system modification | 8
Not completed — Death | 30
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 501
Cronic Heart Failure (CHF) patients with a Cardiac Resynchronization Therapy device system [Number; unit: participants] — Patients with New York Heart Association (NYHA) functional class II-III and severely reduced left ventricular ejection fraction and at least one Heart Failure (HF)-related hospitalisation that required an increase of medication (inotropes, nitrates, diuretics) within the last 12 months were eligible for inclusion. Subject enrolment occurred after successful device implantation (implantable cardioverter-defibrillator (ICD), or a combination of implantable cardiac resynchronization with ICD (CRT-D) and before 34 days post-implant (at time when OptiVol Fluid Trend Data become available).
  participants | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 422
Region of Enrollment [Number; unit: participants]
  Belgium | 44
  United Kingdom | 38
  Germany | 70
  Italy | 115
  France | 58
  Greece | 38
  Israel | 29
  Spain | 23
  Slovakia | 22
  Denmark | 21
  Czech Republic | 19
  Poland | 18
  China | 6
Device therapy [Number; unit: units]
  CRT-D | 393
  ICD | 108

OUTCOME MEASURES:

1. Primary Outcome: Prediction by OptiVol of HF-related Hospitalizations With Signs and/or Symptoms of Pulmonary Congestion.
Time Frame: 34 days post device implant to 6 months
Measure: Number; unit: hospitalization
Groups:
- All Patients: All patients received the same treatment
Arm/Group | All Patients
Number analyzed (Participants) | 501
hospitalization | 58

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 42/501
Other Adverse Events (participants affected / at risk) | 52/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=501)
HF related hospitalization (Cardiac disorders) | 42 (58)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=501)
Heart Failure decompensation (Cardiac disorders) | 52 (104)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No